CLINICAL TRIAL: NCT01219153
Title: Extended High Dose Letrozole Regimen Versus Short Low Dose Letrozole Regimen as an Adjuvant to GnRH Antagonist Protocol in the Management of Patients With Poor Ovarian Response Undergoing IVF-ET, a Randomized Controlled Trial
Brief Title: Extended High Dose Letrozole Regimen Versus Short Low Dose Letrozole Regimen as an Adjuvant to GnRH Antagonist Protocol in the Management of Poor Responders Undergoing IVF-ET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Ahmed Elgazzar Hospital (Other)
Responsible Party: Usama Fouda,M.D, PhD, Cairo university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ext letro/GnRHant
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
Keywords: Letrozole ,IVF, poor responders , GnRH antagonist
MeSH Terms: conditions — Infertility | interventions — LHRH, N-acetyl-(4-chlorophenylalanyl)(1)-(4-chlorophenylalanyl)(2)-tryptophyl(3)-arginyl(6)-alanine(10)-

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended high dose letrozole regimen /GnRH antagonist (Experimental)
  Interventions: Drug: Extended high dose letrozole regimen /GnRH antagonist protocol
- Short low dose letrozole regimen /GnRH antagonist (Active Comparator)
  Interventions: Drug: Short low dose letrozole regimen /GnRH antagonist protocol

INTERVENTIONS:
Drug: Extended high dose letrozole regimen /GnRH antagonist protocol — Letrozole (Femara; Novertis pharma AG, Basle, Switzerland) is administered starting on cycle day one for 8 consecutive days . The dose of letrozole is 5mg /day during the first 5 days of cycle and 2.5 mg/day during the subsequent 3 days .
  Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 5 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Other Names: Extended letrozole/GnRHant
  Arms: Extended high dose letrozole regimen /GnRH antagonist
Drug: Short low dose letrozole regimen /GnRH antagonist protocol — Letrozole (Femara; Novertis pharma AG, Basle, Switzerland)2.5 mg /daily is administered for 5 consecutive days starting on cycle day 3.
  Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 3 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Other Names: Short Letrozole/GnRHant
  Arms: Short low dose letrozole regimen /GnRH antagonist

SUMMARY:
The aim of this randomized controlled trial is to compare the efficacy of extended high dose letrozole regimen (5 mg /day for the first 5 days of cycle and 2.5 mg/day for the subsequent 3 days ) with short low dose letrozole regimen (2,5 mg/day from cycle day 3 to 7 ) as an adjuvant to GnRH antagonist protocol in the management of patients with poor ovarian response undergoing IVF-ET.

DETAILED DESCRIPTION:
Poor response to controlled ovarian stimulation (COH) is estimated to occur in 9-24 % of all IVF cycles. Although there is no consensus on the definition of poor response to COH, inability to produce adequate number of mature follicles( ≤ 2-5) or to recruit adequate number of oocytes ( ≤ 3 oocytes ) in response to standard stimulation protocols are the main criteria used for diagnosis of poor responders .

Patients with poor response to COH usually have higher cyclical cancelation rate , poor embryo quality and less number of embryos suitable for transfer or cryopreservation .

During the past decade gonadotropin releasing hormone antagonists (GnRHant) were widely used in the treatment of patients with poor response to standard gonadotropin releasing hormone agonist (GnRHa) protocols .In contrast to GnRHa, GnRHant is administered at the late follicular phase and therefore don't suppress the early follicular phase endogenous gonadotropins and has no suppressive effect on ovarian function at the stage of follicular recruitment.Several studies comparing GnRHant protocol with the standard GnRHa long protocol revealed a reduction in the duration of stimulation , dose of required gonadotropins , and the costs of IVF cycle with GnRHant as well as equivalent pregnancy rates .

In 2001, Mitwally and Casper introduced letrozole ( a third generation non steroidal aromatase inhibitor licensed for treatment of hormonally-responsive breast cancer after surgery ) as new ovulation induction agent in clomiphene citrate resistant patients with polycystic ovary syndrome (PCOS) . Subsequent studies confirmed the effectiveness of letrozole in induction of ovulation in women with PCOS and in superovulation (either alone or in combination with gonadotropins ) .

In patients with poor response undergoing IVF, several studies revealed that the combination of letrozole ( 2.5 mg or 5 mg/day for 5 consecutive days in early follicular phase ) with GnRHant protocol improved the ovarian response and reduced the gonadotrophin dose required. On the other hand , Schoolcraft et al reported that letrozole(2.5 mg/day from cycle day 3 to 7)/GnRHant protocol has no advantages over microdose flare GnRHa protocol.

The ideal dose and duration of letrozole administration for ovulation and superovulation is still not clear. Several studies comparing two doses of letrozole (2.5 mg or 5 mg) in superovulation suggested that the higher dose might be associated with more follicles developing.

In almost all studies to date , letrozole was administered for five consecutive days in early follicular phase . In only one study , letrozole (2.5 mg/day) was administered for ten consecutive days starting on day 1 of menstrual cycle . In that study , prolonged administration of letrozole produced more mature follicles and pregnancies than short letrozole therapy regimen in patients with clomiphene citrate resistant polycystic ovary syndrome .

The investigators designed this randomized controlled trial to compare the efficacy of extended high dose letrozole regimen (5 mg /day for the first 5 days of cycle and 2.5 mg/day for the subsequent 3 days ) with conventional short low dose letrozole regimen (2,5 mg/day from cycle day 3 to 7 ) as an adjuvant to GnRHant protocol in the management of patients with poor ovarian response undergoing IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

* Patients who produced less than three mature follicles in response to standard GnRH agonist long protocol in their first IVF cycle

Exclusion Criteria:

* Age > 42 years
* FSH> 12 IU/L
* Irregular menstrual cycles
* Unilateral ovary
* Polycystic ovary syndrome
* Endometriosis
* Male factor of infertility requiring ICSI
* History of recurrent miscarriage
* Endocrinologic disorders
* Systemic disease contraindicating pregnancy

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate per started cycle | 5 weeks after embryo transfer
  Presence of intrauterine gestational sac detected by transvaginal ultrasound

SECONDARY OUTCOMES:
Ongoing Pregnancy Rate per started cycle | 18 weeks after embryo transfer
  Pregnancies continued beyond 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D, PhD, Study Chair — Cairo University; Ahmed M Sayed, M.D, PhD, Study Director — Cairo University
Locations (1):
- Ahmed Elgazzar hospital , Assisted conception unit, Giza, Egypt

REFERENCES:
- [Background] Badawy A, Mosbah A, Tharwat A, Eid M. Extended letrozole therapy for ovulation induction in clomiphene-resistant women with polycystic ovary syndrome: a novel protocol. Fertil Steril. 2009 Jul;92(1):236-9. doi: 10.1016/j.fertnstert.2008.04.065. Epub 2008 Aug 15. PMID 18706549
- [Result] Yarali H, Esinler I, Polat M, Bozdag G, Tiras B. Antagonist/letrozole protocol in poor ovarian responders for intracytoplasmic sperm injection: a comparative study with the microdose flare-up protocol. Fertil Steril. 2009 Jul;92(1):231-5. doi: 10.1016/j.fertnstert.2008.04.057. Epub 2008 Aug 3. PMID 18678368
- [Derived] Fouda UM, Sayed AM. Extended high dose letrozole regimen versus short low dose letrozole regimen as an adjuvant to gonadotropin releasing hormone antagonist protocol in poor responders undergoing IVF-ET. Gynecol Endocrinol. 2011 Dec;27(12):1018-22. doi: 10.3109/09513590.2011.579661. Epub 2011 Jun 30. PMID 21714697